CLINICAL TRIAL: NCT04880564
Title: An Open-label, Multi-centre, Phase I/II Study to Investigate the Safety, Tolerability, and Preliminary Efficacy of CN1 in Combination With CN401 in Adult Patients With Relapsed/Refractory Lymphoid Malignancies
Brief Title: A Study of CN1 in Combination With CN401 in Adult Patients With Relapsed/Refractory Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decided that there was no benefit in the drug treatment and due to company change in landscape in the new year.
Sponsor: Curon Biopharmaceutical (Australia) Co Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN1-201
Record Dates: First submitted 2021-04-14; First posted 2021-05-10 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Relapsed Lymphoid Malignancies; Refractory Lymphoid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A (CN1 0.5mg/kg and CN401 400mg) (Experimental): Patients were administered with CN1, 0.5mg/kg, once every three week in combination with 400mg CN401 twice a day, fasted.
  Dosage/Route of admin: CN1- Intravenous Infusion(IV); CN401- Tablet, Oral
  Three to six patients are expected to be enrolled in each arm.
  Interventions: Drug: CN1, 0.5mg/kg and CN401, 400mg
- B (CN1 1mg/kg and CN401 600mg) (Experimental): Patients were administered with CN1, 1mg/kg, once every three week in combination with 600mg CN401 twice a day, fasted.
  Dosage/Route of admin: CN1- Intravenous Infusion(IV); CN401- Tablet, Oral
  Three to six patients are expected to be enrolled in each arm
  Interventions: Drug: CN1, 1mg/kg and CN401, 600mg
- C (CN1 1mg/kg and CN401 800mg) (Experimental): Patients were administered with CN1, 1mg/kg, once every three week in combination with 800mg CN401 twice a day, fasted.
  Dosage/Route of admin: CN1- Intravenous Infusion(IV); CN401- Tablet, Oral
  Three to six patients are expected to be enrolled in each arm
  Interventions: Drug: CN1, 1mg/kg and CN401, 800mg
- D (CN1 3mg/kg and CN401 800mg) (Experimental): Patients were administered with CN1, 3mg/kg, once every three week in combination with 800mg CN401 twice a day, fasted.
  Dosage/Route of admin: CN1- Intravenous Infusion(IV); CN401- Tablet, Oral
  Three to six patients are expected to be enrolled in each arm
  Interventions: Drug: CN1, 3mg/kg and CN401, 800mg
- E (CN1 10mg/kg and CN401 800mg) (Experimental): Patients were administered with CN1, 10mg/kg, once every three week in combination with 800mg CN401 twice a day, fasted.
  Dosage/Route of admin: CN1- Intravenous Infusion(IV); CN401- Tablet, Oral
  Three to six patients are expected to be enrolled in each arm
  Interventions: Drug: CN1, 10mg/kg and CN401, 800mg

INTERVENTIONS:
Drug: CN1, 0.5mg/kg and CN401, 400mg — CN1(0.5mg/kg) will be administered on Day 1 of each cycle (once every three weeks) for up to 12 months and CN401(400mg) will be administered orally twice daily.
  Arms: A (CN1 0.5mg/kg and CN401 400mg)
Drug: CN1, 1mg/kg and CN401, 600mg — CN1(1mg/kg) will be administered on Day 1 of each cycle (once every three weeks) for up to 12 months and CN401(600mg) will be administered orally twice daily.
  Arms: B (CN1 1mg/kg and CN401 600mg)
Drug: CN1, 1mg/kg and CN401, 800mg — CN1(1mg/kg) will be administered on Day 1 of each cycle (once every three weeks) for up to 12 months and CN401(800mg) will be administered orally twice daily.
  Arms: C (CN1 1mg/kg and CN401 800mg)
Drug: CN1, 3mg/kg and CN401, 800mg — CN1(3mg/kg) will be administered on Day 1 of each cycle (once every three weeks) for up to 12 months and CN401(800mg) will be administered orally twice daily.
  Arms: D (CN1 3mg/kg and CN401 800mg)
Drug: CN1, 10mg/kg and CN401, 800mg — CN1(10mg/kg) will be administered on Day 1 of each cycle (once every three weeks) for up to 12 months and CN401(800mg) will be administered orally twice daily.
  Arms: E (CN1 10mg/kg and CN401 800mg)

SUMMARY:
The study is designed to investigate the safety, tolerability and preliminary efficacy in combination with CN1 and CN401 in adult patients with relapsed/refractory lymphoid malignancies.

DETAILED DESCRIPTION:
This is an open-label, multi-center, phase I/II study. The study includes two study drugs CN1 and CN401 and will be conducted in two parts: phase 1 and phase 2.

Phase I: Dose-finding study for the assessment of dose limiting toxicities (DLTs) at 3 or more dose levels in patients with advanced lymphoid malignancies.

Phase II: Expansion study to evaluate the preliminary efficacy of CN1 in combination with CN401 at the RP2D in parallel patient cohorts grouped by non-Hodgkin's Lymphoma (NHL) subtype.

There will 9-18 patients enrolled in the Phase 1 portion of the study and 15- 60 patients will be enrolled in Phase 2 - dosing determined by Phase 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years on the day of signing informed consent.
2. Based on pathology review at the local institution, using the most recent edition of the World Health Organization (WHO) Classification of Tumors of Hematopoietic and Lymphoid Tissues as guidance, leading to the diagnosis of one of the following diseases and their histological subtypes: PTCL, CTCL, and B-cell NHL.
3. Patients must have relapsed or refractory disease after at least one prior systemic anti-tumor treatment.
4. The patients enrolled in Phase II of the study should have received NOT more than five lines of prior systemic therapies.
5. Patients must have at least one evaluable lesion per Lugano 2014 Criteria. Measurable lesions are defined as those that can be accurately measured in at least two dimensions with conventional techniques (positron emission tomography/Computed tomography [PET/CT], magnetic resonance imaging [MRI]) or as > 1.5 cm with spiral CT scan. Patients with non-measurable lesions but assessable diseases (e.g., marrow disease without other radiographically measurable diseases) may be enrolled on a case-by-case basis in discussion with the Sponsor.
6. ECOG performance status 0 to 2.
7. At least 3 months of expected survival.
8. Adequate organ functions, further defined as:

   * Hemoglobin ≥ 9 g/dL.
   * Absolute neutrophil count (ANC) ≥ 1 × 10E+09/L.
   * Platelets ≥ 50 × 10E+09/L (patient without bone marrow [BM] involvement) and ≥ 30 × 10E+09/L (patient with BM involvement).
   * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN if known liver involvement. The ALT and AST should be ≤ 1.5 × ULN in absence of liver involvement/metastasis.
   * Serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance ≥ 50 mL/min (as calculated by the Cockcroft-Gault method).
   * Activated partial thromboplastin time (APTT) or international normalized ratio (INR) ≤ 1.5 × ULN (unless patient is receiving anticoagulants).

Exclusion Criteria:

1. Received any anti-tumour treatment (i.e., chemotherapy, radiotherapy, immunotherapy, biologic therapy, endocrine therapy, etc.,) within four weeks (or five half-lives of the agent, whichever is shorter) prior to the first dose of study drugs, with the following exceptions:

   1. Palliative radiation therapy within 2 weeks.
   2. Oral small molecule targeted therapies within 2 weeks prior to the first dose of study drugs or within 5 half-lives of the drug, whichever is shorter.
   3. Herbal medications within 7 days prior to the first dose.
2. Received other investigational agents (not yet approved by any regulatory agency) within four weeks prior to the first dose of any study drugs.
3. Immunosuppressive medication > 10 mg prednisolone per day or equivalent within 14 days prior to the first dose of the study drug. Note: Use of immunosuppressive medications as prophylaxis in subjects with contrast allergies are acceptable. In addition, temporary uses of corticosteroids considered non-clinically significant may be approved on a case-by-case basis in discussion with the Sponsor.
4. Known clinically active central nervous system (CNS) or meningeal involvement. In the absence of symptoms, investigation into CNS involvement is not required. Patients are eligible if metastases have been treated, patients are neurologically returned to baseline or neurologically stable for at least four weeks and not requiring steroid therapy for at least one week prior to Cycle 1 Day 1.
5. Active infection and in current need of, or likely to need, intravenous (IV) anti-infective therapy.
6. History of immunodeficiency, including history of any positive test result for human immunodeficiency virus (HIV) antibody.
7. Patients who are known to be hepatitis B or C positive (positive HBsAg and/or detectable level of HBV DNA or positive HCV antibody).
8. Active Epstein Barr virus (EBV) unrelated to underlying lymphoma (positive serology for anti-EBV VCA IgM antibody and negative for anti-EBV EBNA IgG antibody, or clinical manifestations and positive EBV polymerase chain reaction [PCR] consistent with active EBV infection).
9. Active CMV (positive serology for anti-CMV IgM antibody, negative for anti-CMV IgG antibody, and positive CMV PCR with clinical manifestations consistent with active CMV infection) and requiring therapy.
10. Current history of a serious uncontrolled medical disorder, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CN1 in combination with CN401 in patients with relapsed/refractory lymphoid malignancies through Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | Measurements at Baseline till completion of last safety visit (270 days)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
To determine maximum tolerated dose and/or Recommended Phase II Dose (RP2D) of CN1 in combination with CN401 | DLT assessed within 21 days after the first dose
  Measured by Incidence of dose limiting toxicities (DLT) during the first cycle of treatment with CN1 in combination with CN401.
To assess the change in anti-tumor activity of CN1 in combination with CN401 through Objective Response Rate analysis | Baseline to End of the Treatment assessed up to an average of 1 year
  Measured/determined by Objective Response Rate

SECONDARY OUTCOMES:
To further evaluate the safety and tolerability of CN1 in combination with CN401 in patients with relapsed/refractory lymphoid malignancies through Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | Measurements at Baseline till completion of last safety visit (270 days)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
To evaluate safety and tolerability of CN1 and CN401 in patients with relapsed/refractory lymphoid malignancies through vital signs as assessed by heart rate | Baseline to End of the Treatment assessed up to an average of 1 year
  Measured by vital sign as assessed by heart rate
To evaluate safety and tolerability of CN1 and CN401 in patients with relapsed/refractory lymphoid malignancies through vital signs as assessed by respiratory rate | Baseline to End of the Treatment assessed up to an average of 1 year
  Measured by vital sign as assessed by respiratory rate
To evaluate safety and tolerability of CN1 and CN401 in patients with relapsed/refractory lymphoid malignancies through vital signs as assessed by body temperature | Baseline to End of the Treatment assessed up to an average of 1 year
  Measured by vital sign as assessed by body temperature
To evaluate safety and tolerability of CN1 and CN401 in patients with relapsed/refractory lymphoid malignancies through vital signs as assessed by pulse, systolic blood pressure, and diastolic blood pressure | Baseline to End of the Treatment assessed up to an average of 1 year
  Measured by vital sign as assessed by pulse, systolic blood pressure, and diastolic blood pressure
To characterize the pharmacokinetics of CN1 and CN401 when administered in combination through Area under the under the drug concentration-time curve. | Baseline to End of the Treatment assessed up to an average of 1 year
  The following parameter is used for evaluation during PK assessments: Area under the drug concentration-time curve (AUC(0-last), AUC0-inf, AUCtau)
To characterize the pharmacokinetics of CN1 and CN401 when administered in combination through Cmax and Tmax. | Baseline to End of the Treatment assessed up to an average of 1 year
  The following parameter is used for evaluation during PK assessments: Maximum concentration (Cmax) and Time to maximum concentration (Tmax)
To characterize the pharmacokinetics of CN1 and CN401 when administered in combination through Apparent terminal half-life (t½). | Baseline to End of the Treatment assessed up to an average of 1 year
  The following parameter is used for evaluation during PK assessments: Apparent terminal half-life (t½)
To characterize the pharmacokinetics of CN1 and CN401 when administered in combination through Apparent terminal elimination rate constant (Kel). | Baseline to End of the Treatment assessed up to an average of 1 year
  The following parameter is used for evaluation during PK assessments: Apparent terminal elimination rate constant (Kel)
To characterize the pharmacokinetics of CN1 and CN401 when administered in combination through Apparent clearance. | Baseline to End of the Treatment assessed up to an average of 1 year
  The following parameter is used for evaluation during PK assessments: Apparent clearance (CL/F and CL/Fss)
To characterize the pharmacokinetics of CN1 and CN401 when administered in combination through Accumulation ration. | Baseline to End of the Treatment assessed up to an average of 1 year
  The following parameter is used for evaluation during PK assessments: Accumulation ration (RA)
To characterize the pharmacokinetics of CN1 and CN401 when administered in combination through Apparent terminal volume of distribution. | Baseline to End of the Treatment assessed up to an average of 1 year
  The following parameter is used for evaluation during PK assessments: Apparent clearance (Vz/F and Vz/Fss)
To further assess change in anti-tumor activity of CN1 in combination with CN401 through ORR | Baseline to End of the treatment visit assessed up to an average of 1 year
  Measured/determined by Objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Jake Shortt, Principal Investigator — Monash Health
Locations (1):
- Monash Health - Monash Medical Centre, Bentleigh, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No